CLINICAL TRIAL: NCT01782664
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Dose Ranging Study to Evaluate the Safety and Efficacy of GSK2586184 in Patients With Chronic Plaque Psoriasis
Brief Title: A Dose Ranging Study to Evaluate the Safety and Efficacy of GSK2586184 in Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116679
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-01

CONDITIONS: Psoriasis
Keywords: PASI; DLQI; GSK2586184; plaque-type psoriasis; PGA; inflammatory gene transcription; JAK-1 inhibitor; serum neopterin; skin biopsy; ACR response criteria; VAS itch score
MeSH Terms: conditions — Psoriasis | interventions — GSK2586184

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 100 mg GSK2586184 (Experimental): Subjects will be randomized to 100 mg GSK2586184 twice daily for up to 84 days
  Interventions: Drug: 100 mg GSK2586184
- 200 mg GSK2586184 (Experimental): Subjects will be randomized to 200 mg GSK2586184 twice daily for up to 84 days
  Interventions: Drug: 200 mg GSK2586184
- 400 mg GSK2586184 (Experimental): Subjects will be randomized to 400 mg GSK2586184 twice daily for up to 84 days
  Interventions: Drug: 400 mg GSK2586184
- Placebo (Placebo Comparator): Subjects will be randomized to receive Placebo twice daily for up to 84 days
  Interventions: Drug: Placebo
- 400 mg GSK2586184 (Cohort B) (Experimental): Subjects will take 400 mg GSK2586184 twice daily for up to 84 days
  Interventions: Drug: 400 mg GSK2586184

INTERVENTIONS:
Drug: 100 mg GSK2586184 — 100 mg GSK2586184 to be taken twice daily with food (as tablets) for up to 84 days.
  Arms: 100 mg GSK2586184
Drug: 200 mg GSK2586184 — 200 mg GSK2586184 to be taken twice daily with food (as tablets) for up to 84 days.
  Arms: 200 mg GSK2586184
Drug: 400 mg GSK2586184 — 400 mg GSK2586184 to be taken twice daily with food (as tablets) for up to 84 days.
  Arms: 400 mg GSK2586184; 400 mg GSK2586184 (Cohort B)
Drug: Placebo — Placebo tablets to be taken twice daily with food for up to 84 days.
  Arms: Placebo

SUMMARY:
A multi-centre, randomised, dose ranging study to evaluate the safety and clinical efficacy of GSK2586184 in patients with chronic plaque psoriasis.

There will be 2 study cohorts (Cohorts A and B). Cohort A is the main study cohort, and this part of the study will be randomised, double-blind and placebo-controlled. Fifty-six subjects will be randomised in Cohort A: 14 subjects in each treatment group: 100 mg, 200 mg or 400 mg GSK2586184, or placebo. Cohort B is an exploratory, open-label investigation of the effect of 400 mg GSK2586184 on inflammatory gene expression in the skin and whole blood, and GSK2586184 concentrations in the skin. A maximum of 8 subjects will be included, and all subjects will take 400 mg GSK2586184.

In both Cohorts A and B, study medication will be administered orally (as tablets), twice daily, for up to 12 weeks.

Each subject will have 7 out-patient visits: Screening; Baseline & Start of treatment; Week 2; Week 4; Week 8; Week 12; and Follow-up (Week 16)

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy subjects with a diagnosis of moderate to severe plaque psoriasis defined by the following criteria:
* Diagnosed for at least 12 months before the first dose of study medication
* Psoriasis plaques cover >=10% of body surface area.
* PASI score of >=12, and PGA score of>=3, and suitable for systemic or light therapy.
* Male or female, between 18 and 75 years of age inclusive.
* Female subjects of childbearing potential must agree to avoid pregnancy and male subjects must agree to avoid female partners becoming pregnant.
* Subjects must agree to use ultra violet (UV) light protection.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Unable to refrain from the use of the following prescription and non-prescription drugs from the following periods before the first dose of study medication until completion of the follow-up visit:
* 12 weeks: alefacept, ustekinumab, adalimumab, etanercept, infliximab, or certolizumab pegol
* 4 weeks or 5 half-lives, whichever is longer:
* systemic medications for other medical conditions that are known to affect psoriasis, including but not limited to oral corticosteroids, cyclosporine, methotrexate, lithium, and beta-adrenergic blockers
* 7 days or 5 half-lives, whichever is longer:
* statins and other OATP and BCRP sensitive substrates (e.g. rapaglinide)
* any agent known to be a substrate of MATE1 and MATE2-K, which undergoes significant renal secretion (e.g. cimetidine)
* 3 weeks or 5 half-lives, whichever is longer:
* any agent known to be a strong CYP3A4 inhibitor or inducer
* 2 weeks: topical therapies that are known to affect psoriasis, including but not limited to corticosteroids, retinoids, vitamin D derivatives, tar and anthralin
* Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis, and will be allowed if in the opinion of the investigator the medication will not interfere with the study procedures or compromise subject safety.
* Phototherapy within 4 weeks before the first dose of study medication.
* A live vaccination within 4 weeks before the first dose of study medication, or a live vaccination planned during the course of the study (until completion of the follow-up visit).
* A major organ transplant (e.g. heart, lung, kidney, liver) or haematopoietic stem cell/marrow transplant.
* Significant unstable or uncontrolled acute or chronic disease unrelated to psoriasis (i.e. cardiovascular including uncontrolled hypertension, hypercholesterolemia, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* A planned surgical procedure that, in the opinion of the investigator, makes the subject unsuitable for the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infections, as follows:
* Known previous or active infection with Mycobacterium Tuberculosis
* Currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
* Hospitalisation for treatment of infection within 60 days before first dose.
* Use of parenteral (IV or intramuscular) antibiotics (antibacterials, antivirals, antifungals, or antiparasitic agents) within 60 days before first dose.
* Unable to refrain from the consumption of grapefruit or grapefruit juice from 3 weeks before the first dose of study medication until 2 weeks after the last dose of study medication.
* History of sensitivity to any components of the study medications, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates their participation.
* Serologic evidence of Hepatitis B (HB) infection based on the results of testing for HBsAg, anti-HBc antibody as follows: subjects positive for HBsAg are excluded; and subjects positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded.
* Positive test for Hepatitis C antibody confirmed sample with a Hepatitis C RIBA immunoblot assay or equivalent. Subjects who are positive for Hepatitis C antibody, but negative when the Hepatitis C RIBA immunoblot assay or equivalent test is performed will be eligible to participate. Subjects who are positive for Hepatitis C antibody and have a positive or indeterminate result when the Hepatitis C RIBA immunoblot assay or equivalent test is performed will not be eligible to participate.
* A positive test for HIV antibody.
* Pregnant females as determined by a positive serum hCG test at screening, or a positive urine hCG test pre-dose on Day 1.
* Lactating females.
* Haemoglobin <11 g/dL, haematocrit <30%, WBC count (absolute) <3 × 10^9/L, neutrophils <1.5 × 10^9/L, platelets <100 × 10^9/L, lymphocytes <1 x 10^9/L.
* Current or history of renal disease, or estimated creatinine clearance <60 mL/min/1.73m^2 or serum creatinine >1.5 ULN.
* Single QTc > 450 msec; or QTc > 480 msec in subjects with Bundle Branch Block.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* ALT > 2xULN; alkaline phosphatase and bilirubin ≥ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within 3 months before the first dose of study medication, or plans to take part in another clinical trial at the same time as participating in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-03-01; Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Germany (8):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- United Kingdom (3):
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, London
  - GSK Investigational Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 68 participants with chronic plaque psoriasis were enrolled. The study was conducted at 13 centers in 2 countries: 10 in Germany and 3 in United Kingdom from 12 March 2013 to 24 March 2014.
Pre-assignment Details: A total of 68 participants were enrolled for this study. Of these, 1 participant was not dosed any study medication because the participant was taking prohibited concomitant medications.
Groups:
- Placebo: Participants received blinded matching placebo orally as tablets, with food, twice daily (BID), for up to 12 weeks.
- GSK2586184 100 mg: Participants received blinded 100 milligrams (mg) GSK2586184 orally as tablets, with food, BID, for up to 12 weeks.
- GSK2586184 200 mg: Participants received blinded 200 mg GSK2586184 orally as tablets, with food, BID, for up to 12 weeks.
- GSK2586184 400 mg: Participants received blinded 400 mg GSK2586184 orally as tablets, with food, BID, for up to 12 weeks.
- GSK2586184 400 mg OL: Participants received Open-Label 400 mg GSK2586184 orally as tablets, with food, BID, for up to 12 weeks.
- GSK2586184 200 mg OL: Participants incorrectly received Open-Label 200 mg (rather than 400 mg) GSK2586184 orally as tablets, with food, BID, for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Started | 14 | 15 | 16 | 14 | 6 | 2
Completed | 8 | 10 | 12 | 9 | 6 | 2
Not Completed | 6 | 5 | 4 | 5 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 2 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL | Total
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.0 (13.79) | 43.9 (14.10) | 49.0 (13.24) | 41.5 (12.08) | 50.7 (11.96) | 53.5 (2.12) | 46.6 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 8 | 3 | 2 | 30
  Male | 9 | 9 | 10 | 6 | 3 | 0 | 37
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Asian - South East Asian Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 14 | 14 | 14 | 14 | 6 | 2 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Achieved >=75% Improvement From Baseline in the Psoriasis Area Severity Index (PASI) Score at Week 12 (PASI 75)
Description: PASI score was determined by evaluation of body surface area (BSA) covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline=Day 1. Percentage of participants who achieved >= 75% improvement from Baseline was reported with last observation carried forward (LOCF) analysis.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Percentage of participants | 0 | 13 | 25 | 57 | 50 | 50

2. Primary Outcome: Percentage of Participants Who Had Achieved >=75% Improvement From Baseline in the Psoriasis Area Severity Index (PASI) Score at Week 12 (PASI 75)
Description: PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline=Day 1. Percentage of participants who achieved >= 75% improvement from Baseline was reported with LOCF analysis.
Time Frame: Baseline and Week 12
Population: Per-Protocol Population: Participants in the ITT analysis set who had no major protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 11 | 14 | 11 | 13 | 4 | 0
Percentage of participants | 0 | 14 | 36 | 62 | 75 |

3. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect. Any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product was recorded from the time a participant consents to participate in the study up to and including any follow-up contact.
Time Frame: From Baseline (Day 1) until the Follow-up visit (Day 112)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Participants
  Any AE | 13 | 10 | 14 | 10 | 6 | 1
  Any SAE | 0 | 2 | 0 | 1 | 1 | 0

4. Secondary Outcome: Number of Participants With the Indicated Hematology Parameters Falling Outside of the Reference Range at Any Time Post-Baseline (BL) During Study
Description: Hematology parameters included: basophils, eosinophils, erythrocyte mean corpuscular hemoglobin (EMCHb) EMCHb concentration (EMCHbC), erythrocyte mean corpuscular volume (EMCV), erythrocyte sedimentation rate (ESR), erythrocytes, hematocrit (fraction 1), hemoglobin, leukocytes, lymphocytes, monocytes, neutrophils, segmented neutrophils, platelets, reticulocytes. BL values were obtained at Day 1. The number of participants with the indicated hematology parameters data outside of the reference range (with high and low) any time post-BL are presented. Anytime post-BL assessments included any scheduled and unscheduled post-BL assessment.
Time Frame: From BL (Day 1) until the Follow-up visit (Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed. Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Participants
  Eosinophils, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Eosinophils, low | 3 | 1 | 0 | 3 | 2 | 0
  Eosinophils, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Eosinophils, high | 0 | 0 | 0 | 2 | 0 | 0
  EMCHbC, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  EMCHbC, low | 6 | 5 | 7 | 5 | 3 | 2
  EMCHb, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  EMCHb, low | 0 | 1 | 1 | 0 | 0 | 0
  EMCHb, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  EMCHb, high | 0 | 1 | 2 | 2 | 3 | 0
  EMCV, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  EMCV, low | 0 | 0 | 1 | 0 | 0 | 0
  EMCV, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  EMCV, high | 0 | 1 | 3 | 2 | 3 | 0
  ESR, high: number analyzed (Participants) | 0 | 0 | 2 | 1 | 2 | 1
  ESR, high |  |  | 1 | 0 | 0 | 1
  Erythrocytes, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Erythrocytes, low | 0 | 1 | 2 | 1 | 0 | 0
  Erythrocytes, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Erythrocytes, high | 1 | 0 | 0 | 0 | 0 | 0
  Hematocrit, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Hematocrit, low | 0 | 0 | 0 | 2 | 0 | 0
  Hematocrit, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Hematocrit, high | 5 | 1 | 4 | 0 | 2 | 0
  Hemoglobin, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Hemoglobin, low | 0 | 2 | 2 | 0 | 0 | 1
  Hemoglobin, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Hemoglobin, high | 1 | 1 | 0 | 1 | 1 | 0
  Leukocytes, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Leukocytes, low | 0 | 2 | 3 | 0 | 0 | 1
  Leukocytes, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Leukocytes, high | 3 | 2 | 4 | 1 | 1 | 0
  Lymphocytes, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Lymphocytes, low | 0 | 0 | 4 | 2 | 0 | 0
  Lymphocytes, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Lymphocytes, high | 0 | 0 | 2 | 0 | 0 | 0
  Monocytes, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Monocytes, low | 2 | 1 | 2 | 3 | 2 | 0
  Monocytes, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Monocytes, high | 1 | 0 | 1 | 0 | 0 | 0
  Neutrophils, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Neutrophils, low | 0 | 1 | 1 | 1 | 0 | 1
  Neutrophils, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Neutrophils, high | 1 | 2 | 3 | 2 | 2 | 0
  Neutrophils, Segmented, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Neutrophils, Segmented, low | 0 | 1 | 1 | 1 | 0 | 1
  Neutrophils, Segmented, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Neutrophils, Segmented, high | 1 | 2 | 3 | 2 | 2 | 0
  Platelets, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Platelets, low | 0 | 1 | 0 | 1 | 0 | 1
  Platelets, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Platelets, high | 1 | 1 | 1 | 0 | 0 | 0
  Reticulocytes, low: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Reticulocytes, low | 3 | 5 | 5 | 4 | 0 | 0
  Reticulocytes, high: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Reticulocytes, high | 2 | 4 | 3 | 1 | 3 | 1

5. Secondary Outcome: Number of Participants With the Indicated Clinical Chemistry Parameters Falling Outside the Reference Range at Any Time Post-Baseline (BL) During the Study
Description: Safety and tolerability were assessed by measuring the clinical chemistry parameters such as creatinine and cystatin C. BL values were obtained at Day 1. The number of participants with the indicated hematology parameter data outside of the reference range (> high or < low) at any time post-BL, including unscheduled or scheduled assessments, are presented.
Time Frame: From Baseline (Day 1) until the Follow-up visit (Day 112)
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Participants
  Creatinine, low, n=13,15,16,14,6,2: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Creatinine, low, n=13,15,16,14,6,2 | 5 | 2 | 4 | 0 | 1 | 0
  Creatinine, high, n=13,15,16,14,6,2: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Creatinine, high, n=13,15,16,14,6,2 | 1 | 0 | 0 | 1 | 0 | 0
  Cystatin C, low, n=13,15,16,14,6,2: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Cystatin C, low, n=13,15,16,14,6,2 | 0 | 0 | 0 | 2 | 0 | 1
  Cystatin C, high, n=13,15,16,14,6,2: number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
  Cystatin C, high, n=13,15,16,14,6,2 | 0 | 0 | 3 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With the Systolic (S) and Diastolic (D) Blood Pressure (BP) Falling Outside the Clinical Concern Range at Any Time Post-baseline During the Study
Description: Vital sign monitoring included systolic and diastolic BP measurements. BP measurements were taken in the supine position after 5 minutes of rest. The number of participants with the SBP or DBP outside the clinical concern range at any time post-BL are presented. SBP "low" was measured as less than 85 millimeters of mercury (mmHg)and "high" was measured as greater than 160 mmHg. DBP "low" was measured as less than 45 mmHg and "high" was measured as greater than 100 mmHg. The BL values were those values obtained at Day 1. Anytime post-BL assessments included any scheduled and unscheduled post-BL assessment.
Time Frame: From Baseline (Day 1) until the follow-up visit (Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
Participants
  SBP, high | 1 | 0 | 0 | 1 | 1 | 0
  DBP, low | 0 | 0 | 0 | 0 | 0 | 0
  DBP, high | 3 | 0 | 0 | 2 | 1 | 0

7. Secondary Outcome: Number of Participants With the Heart Rate Falling Outside the Clinical Concern Range at Any Time Post-Baseline (BL) During the Study
Description: Vital sign monitoring included heart rate (HR) measurements. HR measurements were taken in supine position after 5 minutes of rest. The number of participants with HR outside the clinical concern range at any time post-BL are presented. HR "low" was any HR less than 40 beats per minute (bpm) and "high" was any HR greater than 110 bpm. The BL values were those values obtained at Day 1. Anytime post-BL assessments included any scheduled and unscheduled post-BL assessment.
Time Frame: From Baseline (Day 1) until the Follow-up visit (Day 112)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 13 | 15 | 16 | 14 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 1

8. Secondary Outcome: Change From Baseline in Body Temperature
Description: Vital sign monitoring included body temperature measurements. Body temperature measurements were taken in the supine position after 5 minutes of rest. Baseline is defined as the last result on or before the day of first dose. Change from Baseline was determined by subtracting the indicated time point value minus the Baseline value.
Time Frame: From Baseline (Day 1) until Week 16
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Celsius
  Week 2: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2 | -0.2 (0.54) | -0.0 (0.38) | -0.1 (0.73) | -0.0 (0.36) | 0.0 (0.21) | 0.6 (0.49)
  Week 4: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4 | -0.1 (0.52) | 0.1 (0.44) | -0.1 (0.53) | 0.0 (0.28) | 0.3 (0.37) | 0.0 (0.00)
  Week 8: number analyzed (Participants) | 10 | 12 | 15 | 13 | 6 | 2
  Week 8 | 0.1 (0.44) | 0.1 (0.51) | -0.2 (0.55) | -0.1 (0.28) | 0.2 (0.51) | 0.1 (0.21)
  Week 12: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12 | -0.1 (0.38) | -0.2 (0.64) | -0.1 (0.38) | -0.0 (0.23) | 0.0 (0.29) | 0.2 (0.00)
  Week 16: number analyzed (Participants) | 8 | 10 | 12 | 10 | 6 | 2
  Week 16 | 0.3 (0.45) | -0.1 (0.66) | 0.1 (0.39) | -0.1 (0.21) | 0.4 (0.29) | -0.0 (0.35)

9. Secondary Outcome: Number of Participants With the Indicated Maximum Change From Baseline in the Electrocardiogram (ECG) Findings
Description: ECG measurements were obtained using single 12-lead ECGs with the participant in a supine position after resting in this position for at least 10 minutes. The Baseline values were those values obtained Pre-dose on Day 1. The change from Baseline was the difference between post-Baseline and Baseline. The QT intervals (milliseconds [msec]) corrected for heart rate using Bazett's formula (QTcB) and Fridericia's formula (QTcF) are reported.
Time Frame: From Baseline (Day 1) until the Follow-up visit (Day 112)
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Participants
  QTcB, <30 msec | 13 | 14 | 16 | 12 | 6 | 2
  QTcB, >=30 to <60 msec | 0 | 1 | 0 | 2 | 0 | 0
  QTcF, <30 msec | 13 | 15 | 16 | 12 | 6 | 2
  QTcF, >=30 to <60 msec | 0 | 0 | 0 | 2 | 0 | 0

10. Secondary Outcome: Change From Baseline (BL) in the PASI Score at Week 2, 4, 8 and 12
Description: Psoriatic lesions were assessed using the PASI. PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline=Day 1. The change from Baseline was the difference between post-Baseline and Baseline.
Time Frame: From Baseline (Day 1) until Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Scores on a Scale
  Week 2: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2 | -0.05 (1.716) | -2.39 (3.120) | -0.51 (7.693) | -3.94 (4.766) | -5.25 (4.192) | -3.75 (2.192)
  Week 4: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4 | -0.73 (3.335) | -4.50 (4.344) | -7.03 (7.594) | -8.04 (7.739) | -9.10 (3.854) | -8.20 (0.990)
  Week 8: number analyzed (Participants) | 10 | 12 | 15 | 13 | 6 | 2
  Week 8 | -1.41 (2.122) | -6.54 (6.915) | -8.45 (11.396) | -10.32 (8.293) | -7.85 (5.390) | -11.50 (0.424)
  Week 12: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12 | -3.13 (2.694) | -9.76 (6.341) | -9.21 (12.446) | -13.55 (6.393) | -9.37 (7.181) | -12.45 (1.061)

11. Secondary Outcome: PASI Score at Week 2, 4, 8 and 12
Description: Psoriatic lesions were assessed using the PASI. PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline=Day 1.
Time Frame: Week 2, 4, 8 and 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Scores on a Scale
  Week 2: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2 | 16.33 (4.896) | 16.56 (5.708) | 18.92 (9.969) | 13.39 (5.594) | 13.75 (4.807) | 11.20 (0.283)
  Week 4: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4 | 15.12 (4.683) | 13.94 (6.616) | 12.59 (5.524) | 9.58 (7.910) | 9.90 (6.271) | 6.75 (1.485)
  Week 8: number analyzed (Participants) | 10 | 12 | 15 | 13 | 6 | 2
  Week 8 | 14.64 (4.289) | 12.56 (5.442) | 11.03 (8.322) | 7.30 (9.110) | 11.15 (9.573) | 3.45 (2.899)
  Week 12: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12 | 12.92 (3.384) | 10.52 (4.932) | 9.67 (7.799) | 4.03 (4.666) | 9.63 (10.688) | 2.50 (3.536)

12. Secondary Outcome: Percentage of Participants Who Had a PASI Score With 50%, 75% and 90% Improvement From Baseline Until Week 12
Description: Psoriatic lesions were assessed using the PASI. PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline was Day 1.
Time Frame: From Baseline (Day 1) until Week 12
Population: ITT Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Percentage of Participants
  PASI 50, Week 2 | 0 | 7 | 6 | 7 | 17 | 0
  PASI 50, Week 4 | 0 | 13 | 25 | 57 | 50 | 100
  PASI 50, Week 8 | 0 | 20 | 31 | 71 | 50 | 100
  PASI 50, Week 12 | 0 | 27 | 31 | 64 | 50 | 100
  PASI 75, Week 4 | 0 | 7 | 6 | 21 | 0 | 0
  PASI 75, Week 8 | 0 | 7 | 25 | 50 | 17 | 50
  PASI 75, Week 12 | 0 | 13 | 25 | 57 | 50 | 50
  PASI 90, Week 8 | 0 | 7 | 6 | 14 | 0 | 0
  PASI 90, Week 12 | 0 | 0 | 25 | 36 | 17 | 50

13. Secondary Outcome: Percentage of Participants Who Had a Physician Global Assessment (PGA) Score of 'Clear' (0) or 'Almost Clear' (1) at Weeks 2, 4, 8 and 12
Description: The severity of psoriatic lesions over the whole body were assessed by the investigator using the PGA scoring system. A 0 to 6 point rating scale was used, as follows: 0 = Clear (no signs of psoriasis), 1 = Almost clear (slight elevation, scale and/or erythema), 2 = Mild (mild plaque elevation, scale and/or erythema), 3 = Mild to moderate (mild plaque elevation with moderate erythema and/or scale), 4 = Moderate (moderate plaque elevation, scale and/or erythema), 5 = Moderate to severe (marked plaque elevation, scale and/or erythema), 6 = Severe (very marked plaque elevation, scale and/or erythema). Higher scores indicated worse psoriasis. The Baseline value was the value obtained on Day 1. The scores were reported with the last observation carried forward (LOCF) analysis.
Time Frame: Weeks 2, 4, 8 and 12
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Percentage of Participants
  Week 2 | 0 | 0 | 6 | 0 | 0 | 0
  Week 4 | 0 | 0 | 6 | 0 | 0 | 0
  Week 8 | 0 | 7 | 6 | 29 | 0 | 50
  Week 12 | 0 | 7 | 25 | 43 | 17 | 50

14. Secondary Outcome: Percentage of Participants in Each PGA Score Category at Weeks 2, 4, 8 and 12
Description: as for outcome 13
Time Frame: Weeks 2, 4, 8 and 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Percentage of Participants
  Week 2, Clear: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, Clear | 0 | 0 | 0 | 0 | 0 | 0
  Week 2, almost clear: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, almost clear | 0 | 0 | 6 | 0 | 0 | 0
  Week 2, mild: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, mild | 0 | 0 | 0 | 0 | 0 | 0
  Week 2, mild to moderate: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, mild to moderate | 23 | 14 | 19 | 43 | 33 | 0
  Week 2, moderate: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, moderate | 46 | 64 | 44 | 36 | 50 | 50
  Week 2, moderate to severe: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, moderate to severe | 31 | 14 | 13 | 14 | 0 | 50
  Week 2, severe: number analyzed (Participants) | 13 | 14 | 16 | 14 | 6 | 2
  Week 2, severe | 0 | 7 | 19 | 7 | 17 | 0
  Week 4, Clear: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, Clear | 0 | 0 | 0 | 0 | 0 | 0
  Week 4, almost clear: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, almost clear | 0 | 0 | 7 | 0 | 0 | 0
  Week 4, mild: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, mild | 0 | 14 | 0 | 23 | 33 | 0
  Week 4, mild to moderate: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, mild to moderate | 25 | 36 | 29 | 54 | 33 | 0
  Week 4, moderate: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, moderate | 50 | 29 | 43 | 8 | 17 | 100
  Week 4, moderate to severe: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, moderate to severe | 25 | 14 | 14 | 15 | 17 | 0
  Week 4, severe: number analyzed (Participants) | 12 | 14 | 14 | 13 | 6 | 2
  Week 4, severe | 0 | 7 | 7 | 0 | 0 | 0
  Week 8, Clear: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, Clear | 0 | 0 | 0 | 0 | 0 | 0
  Week 8, almost clear: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, almost clear | 0 | 9 | 7 | 31 | 0 | 50
  Week 8, mild: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, mild | 0 | 9 | 20 | 23 | 50 | 0
  Week 8, mild to moderate: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, mild to moderate | 22 | 27 | 20 | 23 | 17 | 50
  Week 8, moderate,: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, moderate, | 44 | 36 | 33 | 8 | 0 | 0
  Week 8, moderate to severe: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, moderate to severe | 33 | 9 | 13 | 8 | 33 | 0
  Week 8, severe: number analyzed (Participants) | 10 | 11 | 15 | 13 | 6 | 2
  Week 8, severe | 0 | 9 | 7 | 8 | 0 | 0
  Week 12, Clear: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, Clear | 0 | 0 | 7 | 30 | 0 | 50
  Week 12, almost clear: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, almost clear | 0 | 10 | 21 | 20 | 17 | 0
  Week 12, mild: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, mild | 10 | 0 | 0 | 20 | 17 | 0
  Week 12, mild to moderate: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, mild to moderate | 30 | 50 | 29 | 20 | 33 | 50
  Week 12, moderate: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, moderate | 50 | 30 | 21 | 0 | 17 | 0
  Week 12, moderate to severe: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, moderate to severe | 10 | 10 | 21 | 0 | 17 | 0
  Week 12, Severe: number analyzed (Participants) | 10 | 10 | 14 | 10 | 6 | 2
  Week 12, Severe | 0 | 0 | 0 | 10 | 0 | 0

15. Secondary Outcome: Time to PASI 75
Description: PASI 75 was >= 75% improvement from Baseline in PASI score. Psoriatic lesions were assessed by the investigator using a PASI score. PASI score was determined by evaluation of BSA covered by plaque psoriasis in 4 areas (head/neck, arms, trunk and legs with area score of 0.1, 0.2, 0.3 and 0.4 respectively). This test included combination of both degree of involvement (assessed as per the % of affected body area using a 7-point scale such that 0=0% involvement, 1=1-9%, 2=10-29%, 3=30-49%, 4=50-69%, 5=70-89% and 6=90-100%) and severity (evaluated individually using a 5-point scale that ranged as 0=No evidence of sign, 1=slight evidence, 2=moderate evidence, 3=marked evidence and 4=very marked, most severe evidence of sign) of erythema, induration and desquamation in each of the same 4 areas. PASI score ranges from 0(no psoriasis) to 72(worse psoriasis). Final PASI=(sum of severity score for each area)x(% body affected score x area score). Baseline was Day 1.
Time Frame: From Baseline (Day 1) until Week 12
Population: ITT Population. Only participants achieving PASI 75 were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 0 | 2 | 4 | 9 | 3 | 1
Days |  | 59 [33 to 85] | 55.5 [29 to 63] | 57 [27 to 85] | 84 [56 to 85] | 57 [57 to 57]

16. Secondary Outcome: Time to PGA Score of 'Clear' (0) or 'Almost Clear' (1)
Description: The severity of psoriatic lesions over the whole body were assessed by the investigator using the PGA scoring system. A 0 to 6 point rating scale was used, as follows: 0 = Clear (no signs of psoriasis), 1 = Almost clear (slight elevation, scale and/or erythema), 2 = Mild (mild plaque elevation, scale and/or erythema), 3 = Mild to moderate (mild plaque elevation with moderate erythema and/or scale)4 = Moderate (moderate plaque elevation, scale and/or erythema), 5 = Moderate to severe (marked plaque elevation, scale and/or erythema), 6 = Severe (very marked plaque elevation, scale and/or erythema). The Baseline value was the value obtained on Day 1. The scores were reported with the last observation carried forward (LOCF) analysis.
Time Frame: From Baseline (Day 1) until Week 12
Population: ITT Population. Only participants achieving a PGA score of 'Clear' or 'Almost Clear' were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 0 | 1 | 4 | 6 | 1 | 1
Days |  | 55 [55 to 55] | 84.5 [15 to 85] | 57 [55 to 87] | 84 [84 to 84] | 57 [57 to 57]

17. Secondary Outcome: Change From Baseline in the Itch Visual Analogue Scale (VAS) Score at Week 2, 4, 8 and 12
Description: The visual analogue scale (VAS) was used to assess itch. The participants rated the intensity of itch over the past week by marking a line on a 100 millimeter(mm) (0 to 100 mm) long scale. A line placed on the extreme left, that is 0 mm indicated no noticeable itching sensation and extreme right that is 100 mm indicated maximum itching sensation. This scale has no subscales. The participant perception of their symptoms was measured using the VAS itch score. The Baseline value was the value obtained on Day 1. The change from Baseline was the difference between post-Baseline and Baseline.
Time Frame: From Baseline (Day 1) until Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Scores on a Scale
  Week 2: number analyzed (Participants) | 12 | 14 | 15 | 12 | 6 | 2
  Week 2 | -5.67 (32.129) | -14.79 (31.396) | -14.87 (23.670) | -24.92 (24.737) | -56.33 (30.329) | -22.00 (43.841)
  Week 4: number analyzed (Participants) | 10 | 12 | 14 | 12 | 6 | 2
  Week 4 | -7.00 (37.944) | -26.50 (28.659) | -22.36 (27.244) | -28.08 (25.678) | -47.50 (39.480) | -30.00 (62.225)
  Week 8: number analyzed (Participants) | 9 | 11 | 14 | 10 | 6 | 2
  Week 8 | 0.22 (26.138) | -26.27 (35.707) | -24.86 (37.134) | -36.30 (29.788) | -61.50 (31.729) | -32.50 (65.761)
  Week 12: number analyzed (Participants) | 9 | 10 | 13 | 8 | 5 | 2
  Week 12 | -1.56 (34.348) | -21.40 (40.533) | -23.92 (40.586) | -41.13 (31.791) | -60.80 (38.160) | -25.00 (76.368)

18. Secondary Outcome: Itch VAS Scores at Week 2, 4, 8 and 12
Description: The visual analogue scale (VAS) was used to assess itch. The participants rated the intensity of itch over the past week by marking a line on a 100 mm (0 to 100 mm) long scale. A line placed on the extreme left, that is 0 mm indicated no noticeable itching sensation and extreme right that is 100 mm indicated maximum itching sensation. This scale has no subscales. The participant perception of their symptoms was measured using the VAS itch score. Itch VAS scores at Week 2, 4, 8 and 12 are reported.
Time Frame: Week 2, 4, 8 and 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Scores on a Scale
  Week 2,n=12,14,15,12,6,2: number analyzed (Participants) | 12 | 14 | 15 | 12 | 6 | 2
  Week 2,n=12,14,15,12,6,2 | 46.42 (28.909) | 41.64 (21.995) | 42.07 (31.176) | 22.92 (21.707) | 11.83 (14.730) | 42.00 (22.627)
  Week 4,n=10,12,14,13,6,2: number analyzed (Participants) | 10 | 12 | 14 | 13 | 6 | 2
  Week 4,n=10,12,14,13,6,2 | 44.40 (35.485) | 33.42 (25.939) | 32.57 (30.729) | 23.85 (23.140) | 20.67 (30.051) | 34.00 (41.012)
  Week 8,n=9,11,14,11,6,2: number analyzed (Participants) | 9 | 11 | 14 | 11 | 6 | 2
  Week 8,n=9,11,14,11,6,2 | 57.33 (29.368) | 31.55 (29.156) | 29.93 (29.437) | 14.45 (21.920) | 6.67 (7.763) | 31.50 (44.548)
  Week 12,n=9,10,13,9,5,2: number analyzed (Participants) | 9 | 10 | 13 | 9 | 5 | 2
  Week 12,n=9,10,13,9,5,2 | 50.67 (37.683) | 39.50 (33.580) | 30.08 (34.697) | 14.00 (23.701) | 5.40 (6.693) | 39.00 (55.154)

19. Secondary Outcome: Change From Baseline of Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI was used to assess a participant's health-related quality of life. Participants completed the questionnaire to evaluate how their psoriasis affected their life over the week before the assessment took place. Each of the 10 questions was scored out of 0-3 as; 0 = Not at all, 1 = A little, 2 = A lot and 3 = Very much. The total score for the DLQI was calculated by adding up all the individual scores for each question resulting in a minimum of 0 and a maximum of 30. Higher score indicated worsening of participant's quality of life. The Baseline value was the value obtained on Day 1. The change from Baseline was the difference between post-Baseline and Baseline.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants who had a Week 12 evaluation were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 10 | 10 | 14 | 10 | 4 | 2
Scores on a Scale | 1.70 (5.638) | -2.80 (7.743) | -4.29 (8.389) | -8.00 (3.830) | -6.75 (5.123) | -8.00 (11.314)

20. Secondary Outcome: Population Pharmacokinetic (PK) Derived Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the Time of the Last Measureable Concentration (AUC(0-tau) of GSK2586184
Description: Blood samples were taken to measure plasma concentrations of GSK2586184. A two-compartment model with a three-compartment transit model was used to derive PK parameters.
Time Frame: Baseline (pre-dose), Day 14 (2 to 3 hour and 3 to 4 hour post-dose), Day 28 (4 to 6 hour and 6 to 8 hour post-dose), Day 56 (at anytime during clinical visit), Day 84 (1 sample to be taken at anytime during clinical visit)
Population: PK population. The PK Population comprised of all participants who were randomized and received at least one dose of study medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliLitre*hour (ng/mL*hr)
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 0 | 15 | 15 | 14 | 6 | 2
Nanogram/milliLitre*hour (ng/mL*hr) |  | 1464.07903 (43.9) | 3516.96224 (38.7) | 7768.40786 (62.4) | 7561.87974 (79.1) | 3208.20452 (53.5)

21. Secondary Outcome: Clearance of GSK2586184
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)/hr
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 0 | 15 | 15 | 14 | 6 | 2
Litre (L)/hr |  | 68.30232 (43.9) | 56.86726 (38.7) | 51.49060 (62.4) | 52.89690 (79.1) | 62.34017 (53.5)

22. Secondary Outcome: Steady State Volume of Distribution (Vss) of GSK2586184
Description: as for outcome 20
Time Frame: as for outcome 20
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 0 | 15 | 15 | 14 | 6 | 2
L |  | 244.10260 (62.3) | 193.75344 (47.1) | 186.78323 (64.4) | 199.73746 (85.4) | 216.00359 (66.5)

23. Secondary Outcome: Change From Baseline in Serum Neopterin Concentrations at Weeks 2, 4, 8 and 12
Description: Serum Neopterin is a marker of psoriatic disease activity. Blood samples were collected for estimation of serum neoprotein concentration. Baseline was Day 1. The change from Baseline was the difference between post-Baseline and Baseline.
Time Frame: Baseline (pre-dose) and Weeks 2, 4, 8 and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Nanomol per Liter (nmol/L)
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
Number analyzed (Participants) | 14 | 15 | 16 | 14 | 6 | 2
Nanomol per Liter (nmol/L)
  Week 2: number analyzed (Participants) | 13 | 14 | 14 | 12 | 6 | 2
  Week 2 | 0.19 (1.219) | 0.43 (5.394) | 2.35 (6.475) | -0.42 (1.858) | -0.47 (0.918) | 9.95 (13.930)
  Week 4: number analyzed (Participants) | 10 | 14 | 13 | 10 | 6 | 2
  Week 4 | 0.18 (0.844) | -1.69 (2.933) | -1.15 (1.768) | -0.69 (1.195) | -0.67 (0.378) | 1.80 (2.828)
  Week 8: number analyzed (Participants) | 10 | 12 | 15 | 11 | 5 | 2
  Week 8 | -0.14 (0.597) | -1.13 (2.312) | -0.81 (2.294) | 0.31 (2.998) | -0.40 (1.520) | 0.15 (2.192)
  Week 12: number analyzed (Participants) | 8 | 9 | 14 | 9 | 6 | 2
  Week 12 | -0.01 (1.038) | -1.32 (2.355) | -0.79 (1.738) | 4.37 (13.387) | -0.42 (1.182) | 0.35 (0.212)

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events (AEs) were collected from the start of study treatment up to and including the Follow-up visit (up to Study Week 16), Serious AEs were recorded from the time of consent to treatment up to and including the Follow-up visit.
Description: SAEs and non-serious AEs are reported for the Intent-to-Treat Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | GSK2586184 100 mg | GSK2586184 200 mg | GSK2586184 400 mg | GSK2586184 400 mg OL | GSK2586184 200 mg OL
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/16 | 0/14 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/15 | 0/16 | 1/14 | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 13/14 | 10/15 | 14/16 | 10/14 | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | GSK2586184 100 mg (N=15) | GSK2586184 200 mg (N=16) | GSK2586184 400 mg (N=14) | GSK2586184 400 mg OL (N=6) | GSK2586184 200 mg OL (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | GSK2586184 100 mg (N=15) | GSK2586184 200 mg (N=16) | GSK2586184 400 mg (N=14) | GSK2586184 400 mg OL (N=6) | GSK2586184 200 mg OL (N=2)
Nasopharyngitis (Infections and infestations) | 3 | 5 | 4 | 5 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acne pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 5 | 3 | 3 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.